CLINICAL TRIAL: NCT03391791
Title: Long Term Follow-up of Subjects Exposed to Genetically Engineered Tumor Antigen Specific T Cell Receptors
Brief Title: Long Term Follow up of Subjects Exposed to Genetically Engineered T Cell Receptors
Status: Terminated | Type: Observational
Why Stopped: terminated after participants were enrolled
Sponsor: Adaptimmune (Industry)
Responsible Party: Sponsor
Other Study IDs: ADP-0000-003
Record Dates: First submitted 2018-01-02; First posted 2018-01-05 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2018-06

CONDITIONS: Solid and Hematological Malignancies
Keywords: Cell Therapy; T Cell Therapy; SPEAR T Cell; Immuno-oncology; Metastatic; T Cell Receptor; Long Term Follow Up; Genetically Engineered
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genetically engineered T Cell Receptor- treated: Long term follow-up of subjects with solid or hematological malignancies who have received lentivirus-mediated genetically engineered T Cell Receptors in a previous trial
  Interventions: Genetic: Genetically engineered T Cell Receptors

INTERVENTIONS:
Genetic: Genetically engineered T Cell Receptors — No study drug is administered in this study. Subjects who received lentivirus-mediated genetically engineered T Cell Receptors in a previous trial will be evaluated in this trial for long-term safety and efficacy.

SUMMARY:
Subjects who previously took part in an Adaptimmune study and received genetically changed T cells (including but not limited to MAGE-A10ᶜ⁷⁹⁶T and MAGE-A4ᶜ¹º³²T) are asked to take part in this long term follow-up study. Subjects will be asked to join this study once they complete the parent interventional study.

The purpose of this study is to find out if the genetically changed T cells that subjects received in the parent study have any long-term side effects. No additional study drug will be given, but subjects can receive other therapies for their cancer while they are being followed for long term safety in this study.

For a period of 15 years starting from last administration of the genetically changed T cells, subjects will visit their study doctor for a check-up and to have blood tests to look for any changes that might have happened because of the genetically changed T cells.

DETAILED DESCRIPTION:
This is a non-therapeutic, multi-center, long-term follow-up (LTFU) study of subjects who have received lentivirus-mediated genetically engineered T Cell Receptors in an Adaptimmune sponsored clinical trial. The study is designed in accordance with FDA and EMA guidance on gene therapy trials.

The study involves up to 15 years post-infusion monitoring of subjects who have been exposed to lentivirus-mediated gene transfer in Adaptimmune clinical studies. The study will include subjects who have received various T cell receptors including but not limited to MAGE-A10ᶜ⁷⁹⁶T and MAGE-A4ᶜ¹º³²T. Subjects will undergo clinical evaluation (i.e., new medical history, physical exam, adverse events, and exposure to mutagenic agents, anti-cancer therapies and investigational products in other clinical studies) with careful attention to adverse events possibly related to gene transfer or lentivirus-induced diseases. Blood samples will be collected for evaluating persistence of cells with lentiviral vector sequences, the detection of replication competent lentivirus (RCL), and chemistry and hematology laboratory assessments. Subjects will be followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have received T cell receptor therapy in an Adaptimmune clinical study
* Subjects who have provided informed consent prior to their study participation

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with solid or hematological malignancies rolling over from interventional study where they were treated with a genetically modified T-cell receptor
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

PRIMARY OUTCOMES:
Number of subjects with specific Long Term Follow-Up adverse events (AEs), including serious adverse events (SAEs) associated with administration of autologous T cell receptors that have been genetically modified by lentiviral vectors. | 15 years post last treatment
  * New malignancies
  * New incidence or exacerbation of a pre-existing neurologic disorder
  * New incidence or exacerbation of a prior rheumatologic or other autoimmune disorder
  * New incidence of a hematologic disorder
  * Opportunistic and/or serious infections
  * Unanticipated illness and/or hospitalization deemed related to gene modified cell therapy

SECONDARY OUTCOMES:
Measurement of Replication Competent Lentivirus (RCL) in genetically modified T cells | 15 years post last treatment
  Subjects' peripheral blood samples will be used to evaluate RCL
Persistence of genetically modified cells in the body | 15 years post last treatment
  Peripheral blood samples will be used to evaluate persistence
Assess the pattern of vector integration sites if at least 1% of cells in the surrogate sample are positive for vector sequences by PCR | 15 years post last treatment
  Number of samples positive for vector integration by PCR
Overall Survival (OS) post-infusion | 15 years post last treatment
  OS defined as the interval between the date of first T cell infusion and date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Butler, MD, Principal Investigator — Princess Margaret Cancer Centr
Locations (3):
- United States (2):
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Cancer Centr, Toronto, Ontario, Canada